CLINICAL TRIAL: NCT04398615
Title: Validazione Dell'Orologio ADAMO Per l'Individuazione Precoce Delle Cadute Nel Paziente Anziano
Brief Title: Validation of the ADAMO Watch for the Early Detection of Fall Events in Older Patients
Acronym: ADAMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: Caretek S.r.l. Turin, Italy (Unknown); Consoft Sistemi S.p.A. Turin, Italy (Unknown)
Responsible Party: Principal Investigator, Dott.ssa RENATA MARINELLO, Principal Investigator, A.O.U. Città della Salute e della Scienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ADAMO
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Accidental Falls; Wearable Electronic Devices
Keywords: Aged; Telemetry; Wearable Electronic Devices; Fall detection

STUDY DESIGN:
Masking Description: During the follow-up period both healthcare personnel and investigators will not be aware of data (including fall events) registered by the experimental device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Single arm, receiving the experimental device
  Interventions: Device: Wearable watch device

INTERVENTIONS:
Device: Wearable watch device — Every study participant will be given a wearable watch device at the beginning of the study and will be instructed on how to use the device and to wear it continuously throughout the duration of the study (6 months total follow-up). The device will register biometric data and automatically archived. During the follow-up period both healthcare personnel and investigators will not be aware of data (including fall events) registered by the experimental device.
  Other Names: ADAMO

SUMMARY:
"La Casa nel Parco" (CANP) Project is a multidisciplinary project funded by the European Union and Regione Piemonte aimed to explore innovative technology application in the care of older subjects. In this context, ADAMO is a single arm open label trial evaluating the capability of a wearable watch device to correctly detect fall events in community-dwelling older subjects aged 75 years and older, at high risk of falls. Secondary objectives of the study are to identify specific patterns on telemetric measures and health status variations able to predict future fall events, and to evaluate the tolerability and the influence on patient's quality of life of this wearable device.

The main objectives of the study are to evaluate the impact of the intervention on 1) medication adherence after discharge 2) medication appropriateness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 years and older
* At least 2 fall events during the 12 months previous to enrollment
* Signed written informed consent

Exclusion Criteria:

* Severe cognitive impairment
* Bedridden condition
* Patients unable to walk autonomously (walking aids allowed)

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of self-reported fall events | 6 months
  Fall event incidence evaluated through scheduled phone call interviews with the patient or the caregiver, from enrollment every 15 days through to 6 months, recording also timing and context of event, environmental factors, health status at the moment of the event, health consequences, therapeutic modifications.
Incidence of device-reported fall events | 6 months
  Fall event incidence automatically evaluated by the wearable watch device, based on biometric data continuously recorded from enrollment through to 6 months.

SECONDARY OUTCOMES:
Variation in quality of life reported at three levels EQ-5D (EQ-5D-5L) Questionnaire | At enrollment and at 6 months
  Patient's quality of life will be evaluated both at enrollment and at 6 months through the five levels EQ-5D (EQ-5D-3L) Questionnaire, exploring the five dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety depression (each dimension scored 1-3, with 3 indicating worse problems), and a general measure of perceived health on a Visual Analogue Scale (EQ-VAS), scored 0-100 (with 100 indicating the best perceived health possible)
Variation in fear of falling evaluated with Short Falls Efficacy Scale International (Short FES-I) | At enrollment and at 6 months
  Patient's fear of falling be evaluated both at enrollment and at 6 months through the Short Falls Efficacy Scale International (Short FES-I) Status (minimum 7-maximum 28, higher levels indicating most severe concern about falling)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Marinello, MD, PhD, Principal Investigator — OAU Città della Salute e della Scienza di Torino, Turin, Italy
Locations (1):
- S.C. Geriatria e Malattie Metaboliche dell'Osso U, A.O.U. Città della Salute e della Scienza di Torino, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheffer AC, Schuurmans MJ, van Dijk N, van der Hooft T, de Rooij SE. Fear of falling: measurement strategy, prevalence, risk factors and consequences among older persons. Age Ageing. 2008 Jan;37(1):19-24. doi: 10.1093/ageing/afm169. PMID 18194967
- [Background] Kempen GI, Yardley L, van Haastregt JC, Zijlstra GA, Beyer N, Hauer K, Todd C. The Short FES-I: a shortened version of the falls efficacy scale-international to assess fear of falling. Age Ageing. 2008 Jan;37(1):45-50. doi: 10.1093/ageing/afm157. Epub 2007 Nov 20. PMID 18032400
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Ganz DA, Higashi T, Rubenstein LZ. Monitoring falls in cohort studies of community-dwelling older people: effect of the recall interval. J Am Geriatr Soc. 2005 Dec;53(12):2190-4. doi: 10.1111/j.1532-5415.2005.00509.x. PMID 16398908
- See also: EuroQol EQ-5D — http://www.euroqol.org/.